CLINICAL TRIAL: NCT04051372
Title: Diagnosis of Lung Complication After Allogeneic Hematopoietic Stem Cell Transplantation by Multiple Parameter System Through Bronchoscopic Alveolar Lavage
Brief Title: Diagnosis of Lung Complication After Allo-HSCT by Multiple Parameter System Through BAL
Acronym: SHSYXY-BAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 2018KY270
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Bronchoalveolar Lavage Fluid; Lung Infection
Keywords: Idiopathic Pneumonia Syndrome; CMV Pneumonia; Pneumocystis Jiroveci Pneumonia; Invasive Pulmonary Aspergillosis
MeSH Terms: conditions — Pneumonia, Pneumocystis; Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAL group: Adult patients with hematology disease under allo-HSCT at any phase of treatment are enrolled according to the following criteria:
  1. lung infiltration detection at computed tomography (CT) scan.
  2. Patients with fever, cough, respiratory symptoms. According to the investigators, the patients fulfilling these criteria undergo BAL as soon as possible
  Interventions: Diagnostic Test: Bronchoscopic Alveolar Lavage

INTERVENTIONS:
Diagnostic Test: Bronchoscopic Alveolar Lavage — The diagnostic yield of different diagnostic methods for lung infection and non-infectious diseases under allo-HSCT patients.
  1. Classic microbiological cultures designed for bacteria, fungi, and mycobacteria.
  2. Detection of human cytomegalovirus (CMV) and EB virus in serum and BAL was tested using a Real-time PCR kit.
  3. Detection of aspergillus galactomannan antigen 1,3-beta-D-glucan in serum and BAL was performed using an enzyme immunoassay method.
  4. Cytological and pathogenic microscopic evaluation in BALF
  5. Flow cytological analysis of T lymphocyte subsets in BALF and serum
  6. Cytokine detection in BALF and serum
  7. Microbiology detection in BALF by mNGS

SUMMARY:
The aim of this study was to evaluate the diagnostic yield for lung complication after allo-HSCT by multiple parameter system through BAL.

DETAILED DESCRIPTION:
一) Adult patients with hematology disease under allo-HSCT at any phase of treatment are enrolled according to the following criteria:

1. lung infiltration detection at computed tomography (CT) scan.
2. Patients with fever, cough, respiratory symptoms. According to the investigators, the patients fulfilling these criteria undergo BAL as soon as possible

二) The BALF samples were tested using such methods

1. classic microbiological cultures designed for bacteria, fungi, and mycobacteria.
2. Detection of human cytomegalovirus (CMV) and EB virus in serum and BAL was tested using a Real-time PCR kit.
3. Detection of aspergillus galactomannan antigen 1,3-beta-D-glucan in serum and BAL was performed using an enzyme immunoassay method.
4. Cytological and pathogenic microscopic evaluation in BALF
5. Flow cytological analysis of T lymphocyte subsets in BALF and serum
6. Cytokine detection in BALF and serum
7. Microbiology detection in BALF by mNGS

三) Pathogenic spectrum analysis and Targeted etiological therapy

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hematological diseases.
2. Recipients of allogeneic peripheral blood stem cell transplantation.
3. Lung infiltration detection at computed tomography (CT) scan.
4. Patients with fever, cough, respiratory symptoms.
5. Consent to BAL and follow-up observation after BAL

Exclusion Criteria:

1. Severe bleeding tendency, platelet less than 20000/uL, or severe coagulation dysfunction;
2. Multiple bullae are at risk of rupture;
3. Untreated patients with active pulmonary tuberculosis;
4. Patients with severe consumptive diseases or conditions and various causes can not cooperate well
5. Cardiac insufficiency, severe pulmonary ventilation dysfunction
6. Recent massive hemoptysis
7. Aortic aneurysm and esophageal varices are at risk of rupture

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High morbidity and mortality in patient receiving hematopoietic Stem Cell Transplantation (HSCT) are resulted from lung complications. Diagnosis of the etiology affects the choice of treatment. The bronchoalveolar lavage (BAL) analysis is safe and widely accepted, which provide valuable information for pathogen identification in pulmonary infections diagnosis.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 100 days after BAL
  Efficiency of treatment for pulmonary complications after allo-HSCT

SECONDARY OUTCOMES:
microbiology diagnostic yields | 100 days after BAL
  Comparing the pathogenic detection rate by BALF with non-invasive detection method
all-cause mortality and attributable mortality of pulmonary complications | 30-day and 100-day after BAL
  30-day and 100-day mortality (including all-cause mortality and attributable mortality of pulmonary complications) in patients undergoing BAL

CONTACTS AND LOCATIONS:
Overall Officials: xianmin song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

REFERENCES:
- [Derived] Shen Z, Wang Y, Bao A, Yang J, Sun X, Cai Y, Wan L, Huang C, Xu X, Niu J, Xia X, Shen C, Wei Y, Qiu H, Zhou K, Zhang M, Tong Y, Song X. Metagenomic Next-Generation Sequencing for Pathogens in Bronchoalveolar Lavage Fluid Improves the Survival of Patients with Pulmonary Complications After Allogeneic Hematopoietic Stem Cell Transplantation. Infect Dis Ther. 2023 Aug;12(8):2103-2115. doi: 10.1007/s40121-023-00850-w. Epub 2023 Aug 4. PMID 37541984